CLINICAL TRIAL: NCT02959086
Title: Shanghai Epidemiology Study for Adolescents and Children with Cancer
Status: Recruiting | Type: Observational
Sponsor: Children's Cancer Group, China (Network)
Collaborators: Shanghai Children's Medical Center (Other); Shanghai Municipal Center for Disease Prevention & Control (Unknown)
Responsible Party: Sponsor
Other Study IDs: CCGChina
Record Dates: First submitted 2016-11-07; First posted 2016-11-08 (Estimated); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Childhood Cancer
Keywords: Epidemiology; Shanghai; Cancer; Adolescents; Children
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Patients were diagnosed since January 2002.

SUMMARY:
The purpose of this study is to describe the morbidity, mortality, disability and survival rate in Shanghai adolescents and children with cancer diagnosed since January 2002.

DETAILED DESCRIPTION:
The investigators collected information of all the adolescents and children diagnosed cancer in Shanghai since January 2002, including their name, gender, the date of birth, the diagnosis date, disease diagnosis, residence address and the last follow-up time status (survival/death). The type of cancer included all malignant tumors such as Acute Lymphocytic Leukemia, Acute Myeloid Leukemia, Non-Hodgkin Lymphoma, Hodgkin Lymphoma, central nervous system tumors, Neuroblastoma, Wilms tumor and so on. Then the investigators would analyze the morbidity, mortality, disability and survival rate.

ELIGIBILITY:
Inclusion Criteria:

* 0-19 year-old children and adolescents.
* Diagnosed cancer in Shanghai since January 2002.

Exclusion Criteria:

* Patients who were lost of follow-up.
* Patient's death wasn't caused by cancer or complications but by other accidents such as car accident, fell from a great height and so on.

Ages: 0 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Since January 2002 in Shanghai, 0-19 year-old children and adolescents diagnosed with cancer.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2002-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival for the whole cohort | 5 years

SECONDARY OUTCOMES:
Mortality for the whole cohort | 5 years

OTHER OUTCOMES:
Disability rate for the whole cohort | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Jin Gao, MD, Principal Investigator — Shanghai Children's Medical Center
Locations (2):
- China (2):
  - Shanghai Children's Medical Center, Shanghai, Shanghai Municipality
  - Shanghai Municipal Center of Disease Prevention & Control, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No